CLINICAL TRIAL: NCT00913952
Title: Comparative, Randomized, 3-way Crossover Bioavailability Study of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules In Health Adult Males Under Fed and Fasted Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 940155
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Depression
Keywords: Antidepressant
MeSH Terms: conditions — Depression | interventions — Clomipramine

ARMS (3):
- 1 (Experimental): Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fasting Conditions.
  Interventions: Drug: Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fasting Conditions
- 2 (Experimental): Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions.
  Interventions: Drug: Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions
- 3 (Active Comparator): Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions.
  Interventions: Drug: Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions

INTERVENTIONS:
Drug: Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fasting Conditions
  Arms: 1
Drug: Geneva 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions
  Arms: 2
Drug: Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules Under Fed Conditions
  Arms: 3

SUMMARY:
To demonstrate the relative bioavailability of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride capsules under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1994-04; Primary Completion 1994-06 (Actual); Study Completion 1994-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 53 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lalonde, Pharm.D., Principal Investigator — Phoenix International Life Science Inc.